CLINICAL TRIAL: NCT00418834
Title: A Multicenter, Randomized, Double-Blind, Parallel Arm, 12-Week Study to Evaluate the Efficacy and Safety of Ezetimibe 10 mg When Added to Atorvastatin 10 mg Versus Titration to Atorvastatin 20 mg and to 40 mg in Elderly Patients With Hypercholesterolemia at High Risk for CHD
Brief Title: Ezetimibe and Atorvastatin vs. Atorvastatin in Patients Age 65 and Older at High Risk for Coronary Heart Disease (CHD)(0653-112)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653-112; MK0653-112; 2006_549
Record Dates: First submitted 2007-01-03; First posted 2007-01-05 (Estimated); Results first posted 2009-10-06 (Estimated); Last update posted 2024-05-14 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: ezetimibe and atorvastatin; Drug: Placebo (unspecified)
- 2 (Active Comparator)
  Interventions: Drug: atorvastatin; Drug: Placebo (unspecified)

INTERVENTIONS:
Drug: ezetimibe and atorvastatin — ezetimibe 10 mg and atorvastatin 10 mg daily for 12 weeks
  Arms: 1
Drug: atorvastatin — Atorvastatin 20 mg daily for 6 weeks, and up-titrated to atorvastatin 40 mg daily for an additional 6 weeks
  Arms: 2
Drug: Placebo (unspecified) — Placebo (unspecified) daily for 12 weeks

SUMMARY:
A 12 week clinical trial in patients 65 years of age and older with hypercholesterolemia at high risk for coronary heart disease to study the effects of atorvastatin and ezetimibe given in combination and two higher doses of atorvastatin on lipid lowering.

ELIGIBILITY:
Inclusion Criteria:

* Patient is age 65 or older
* Patient is willing to maintain cholesterol lowering diet
* Patient has hyperlipidemia with LDL level greater than 70 mg/dl or 100 mg/dl depending on their CHD risk category

Exclusion Criteria:

* A condition which, in the opinion of the investigator, would pose a risk to the patient or interfere with participation in the study
* Patient is unlikely to be compliant in taking study medication
* Patient with chronic or unstable medical condition
* Patient is taking unstable doses of medication
* Patient drinks more than 2 alcoholic drinks per day
* Patient has elevations in certain laboratory values (CK, AST, ALT)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1053 (Actual)
Dates: Start 2007-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zieve F, Wenger NK, Ben-Yehuda O, Constance C, Bird S, Lee R, Hanson ME, Jones-Burton C, Tershakovec AM. Safety and efficacy of ezetimibe added to atorvastatin versus up titration of atorvastatin to 40 mg in Patients > or = 65 years of age (from the ZETia in the ELDerly [ZETELD] study). Am J Cardiol. 2010 Mar 1;105(5):656-63. doi: 10.1016/j.amjcard.2009.10.029. Epub 2009 Dec 24. PMID 20185012
- [Derived] Constance C, Ben-Yehuda O, Wenger NK, Zieve F, Lin J, Hanson ME, Lowe RS, Tershakovec AM. Atorvastatin 10 mg plus ezetimibe versus titration to atorvastatin 40 mg: attainment of European and Canadian guideline lipid targets in high-risk subjects >/=65 years. Lipids Health Dis. 2014 Jan 13;13:13. doi: 10.1186/1476-511X-13-13. PMID 24411003

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase III
  First Patient In: 28-Feb-2007; Last Patient Last Visit: 01-Oct-2008
  143 centers worldwide (United States, Canada, Poland, Romania, Ukraine and Russia)
Pre-assignment Details: Patients were stratified based on baseline LDL-C levels and presence or absence of atherosclerotic vascular
  disease to achieve balance across treatment groups.
Groups:
- Atorva 10 mg + EZ: [Atorva 10 mg + Ezetimibe 10 mg] orally once daily for 12 weeks
- Atorva 20 mg / Atorva 40 mg: Atorva 20 mg orally once daily for 6 weeks, and up-titrated to Atorva 40 mg orally once daily for an additional 6 weeks
Period: Overall Study
Arm/Group | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg
Started | 526 | 527
Completed | 503 | 507
Not Completed | 23 | 20
Not completed — Adverse Event | 16 | 9
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 4 | 3
Not completed — Withdrawal by Subject | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg | Total
Number analyzed (Participants) | 526 | 527 | 1053
Age, Continuous [Mean (Full Range); unit: years] | 71.2 [65 to 86] | 71.2 [65 to 92] | 71.2 [65 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 277 | 286 | 563
  Male | 249 | 241 | 490
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 503 | 505 | 1008
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Asian | 2 | 3 | 5
  Black | 21 | 17 | 38
  Multi-Racial | 0 | 1 | 1
Region of Enrollment [Number; unit: Participants]
  North America | 189 | 197 | 386
  Europe | 337 | 330 | 667
BMI [Body Mass Index (<30, ≥30 kg/m2)] [Number; unit: Participants]
  <30 kg/m2 | 359 | 362 | 721
  ≥30 kg/m2 | 165 | 165 | 330
  Missing | 2 | 0 | 2
Apo lipoprotein A-I (Apo A-I) [Mean (Standard Deviation); unit: mg/dL] | 164.3 (28.7) | 164.4 (26.8) | 164.4 (27.7)
Apo lipoprotein B (Apo B) [Mean (Standard Deviation); unit: mg/dL] | 103.6 (22.8) | 101.8 (21.4) | 102.7 (22.1)
Apo lipoprotein B (Apo B):Apo lipoprotein A-I (Apo A-I) Ratio [Mean (Standard Deviation); unit: Ratio] | 0.6 (0.2) | 0.6 (0.2) | 0.6 (0.2)
High Density Lipoprotein Cholesterol (HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 54.9 (13.6) | 54.5 (12.3) | 54.7 (13.0)
Highly selective C-reactive protein (hs-CRP) [Mean (Standard Deviation); unit: mg/L] — Robust Standard Deviation was calculated for hs-CRP as: interquartile range
  (IQR)/1.075, where IQR=3rd quartile - 1st quartile.
  mg/L | 1.8 (2.7) | 1.9 (2.3) | 1.9 (2.5)
Low Density Lipoprotein Cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] | 102.9 (27.7) | 101.8 (20.7) | 102.3 (24.4)
Low Density Lipoprotein Cholesterol (LDL-C):High Density Lipoprotein Cholesterol (HDL-C) Ratio [Mean (Standard Deviation); unit: Ratio] | 2.0 (0.7) | 2.0 (0.6) | 2.0 (0.7)
Non-High Density Lipoprotein Cholesterol (Non-HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 128.2 (30.6) | 127.2 (25.2) | 127.7 (28.1)
Non-High Density Lipoprotein Cholesterol (Non-HDL-C):High Density Lipoprotein Cholesterol (HDL-C) Ra [Mean (Standard Deviation); unit: Ratio] | 2.5 (0.9) | 2.5 (0.8) | 2.5 (0.9)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 183.1 (31.8) | 181.8 (26.1) | 182.4 (29.1)
Total Cholesterol (TC):High Density Lipoprotein-C (HDL-C) Ratio [Mean (Standard Deviation); unit: Ratio] | 3.5 (0.9) | 3.5 (0.8) | 3.5 (0.9)
Triglycerides (TG) [Mean (Standard Deviation); unit: mg/dL] — Robust Standard Deviation was calculated for Triglycerides as: interquartile range (IQR)/1.075, where IQR=3rd quartile - 1st quartile.
  mg/dL | 112.8 (55.3) | 116.5 (60.0) | 114.0 (56.7)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in LDL-C at Week 6
Time Frame: Baseline and Week 6
Population: Full Analysis Set (FAS): The FAS population
  includes all randomized patients who took at least 1 dose of study medication and had a baseline (BL) value and at
  least one post BL value. Post BL measurements up to 3 days following the last dose of double-blind study medication
  were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg
Number analyzed (Participants) | 515 | 515
Percent Change | -26.7 [-28.6 to -24.7] | -12.8 [-14.8 to -10.9]
Statistical Analysis 1: Comparison: Atorva 10 mg + EZ vs Atorva 20 mg / Atorva 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, baseline LDL-C, and AVD status; Mean Difference (Final Values) = -13.8, 95% CI [-16.0 to -11.7], Standard Error of Mean 1.1 — (Atorva 10 mg + EZ minus Atorva 20 mg)

2. Secondary Outcome: Percent Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C) at Week 12
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg
Number analyzed (Participants) | 516 | 509
Percent Change | -22.5 [-25.0 to -19.9] | -17.9 [-20.5 to -15.4]
Statistical Analysis 1: Comparison: Atorva 10 mg + EZ vs Atorva 20 mg / Atorva 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, baseline LDL-C, and AVD status; Mean Difference (Final Values) = -4.6, 95% CI [-7.4 to -1.8], Standard Error of Mean 1.4 — (Atorva 10 mg + EZ minus Atorva 20 mg)

3. Secondary Outcome: Number of Patients Who Achieved Low Density Lipoprotein Cholesterol (LDL-C) <70 mg/dL at Week 6
Time Frame: Week 6
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg
Number analyzed (Participants) | 515 | 515
Participants
  <70 mg/dL | 244 | 92
  ≥70 mg/dL | 271 | 423
Statistical Analysis 1: Comparison: Atorva 10 mg + EZ vs Atorva 20 mg / Atorva 40 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Model terms: treatment, baseline LDL-C, and AVD status; Odds Ratio (OR) = 6.32, 95% CI [4.52 to 8.84] — Estimated ratio is the predictive odds of attaining LDL-C target on Atorva 10 mg + EZ versus Atorva 20 mg

4. Secondary Outcome: Number of Patients Who Achieved Low Density Lipoprotein Cholesterol (LDL-C) <70 mg/dL at Week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg
Number analyzed (Participants) | 516 | 509
Participants
  <70 mg/dL | 225 | 164
  ≥70 mg/dL | 291 | 345
Statistical Analysis 1: Comparison: Atorva 10 mg + EZ vs Atorva 20 mg / Atorva 40 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Model terms: treatment, baseline LDL-C, and AVD status; Odds Ratio (OR) = 1.87, 95% CI [1.40 to 2.50] — Estimated ratio is the predictive odds of attaining LDL-C target on Atorva 10 mg + EZ versus Atorva 20 mg / Atorva 40 mg

5. Secondary Outcome: Number of Patients Who Achieved LDL-C <100 mg/dL for Patients Without Atherosclerotic Vascular Disease (AVD) and LDL-C <70 mg/dL for Patients With Atherosclerotic Vascular Disease (AVD) at Week 6
Time Frame: Week 6
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg
Number analyzed (Participants) | 515 | 515
Participants
  <100 mg/dL (w/o AVD) and <70 mg/dL (w/ AVD) | 274 | 127
  >100 mg/dL (w/o AVD) and ≥70 mg/dL (w/AVD) | 241 | 388
Statistical Analysis 1: Comparison: Atorva 10 mg + EZ vs Atorva 20 mg / Atorva 40 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Model terms: treatment, baseline LDL-C, and AVD status; Odds Ratio (OR) = 5.48, 95% CI [3.98 to 7.55] — Estimated ratio is the predictive odds of attaining LDL-C target on Atorva 10 mg + EZ versus Atorva 20 mg

6. Secondary Outcome: Number of Patients Who Achieved LDL-C<100 mg/dL for Patients Without AVD and LDL-C<70 mg/dL for Patients With AVD at Week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg
Number analyzed (Participants) | 516 | 509
Participants
  <100 mg/dL (w/o AVD) and <70 mg/dL (w/ AVD) | 255 | 200
  ≥100 mg/dL (w/o AVD) and ≥70 mg/dL (w/ AVD) | 261 | 309
Statistical Analysis 1: Comparison: Atorva 10 mg + EZ vs Atorva 20 mg / Atorva 40 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Model terms: treatment, baseline LDL-C, and AVD status; Odds Ratio (OR) = 1.75, 95% CI [1.32 to 2.31] — [estimate comment as in outcome 4, analysis 1]

7. Other Pre Specified Outcome: Percent Change From Baseline in High Density Lipoprotein Cholesterol (HDL-C) at Week 6
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg
Number analyzed (Participants) | 515 | 515
Percent Change | 2.5 [1.1 to 4.0] | 0.7 [-0.8 to 2.1]
Statistical Analysis 1: Comparison: Atorva 10 mg + EZ vs Atorva 20 mg / Atorva 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, baseline HDL-C, and AVD status; Mean Difference (Final Values) = 1.9, 95% CI [0.3 to 3.5], Standard Error of Mean 0.8 — (Atorva 10 mg + EZ minus Atorva 20 mg)

8. Other Pre Specified Outcome: Percent Change From Baseline in High Density Lipoprotein Cholesterol (HDL-C) at Week 12
Time Frame: Baseline and Week 12
Population: Full Analysis Set (FAS): The FAS population includes all randomized patients who took at least 1 dose of study medication and had a baseline (BL)value and at least one post BL value. Post BL measurements up to 3 days following the last dose of double-blind study medication were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg
Number analyzed (Participants) | 516 | 509
Percent Change | 2.4 [0.9 to 3.8] | -0.8 [-2.2 to 0.7]
Statistical Analysis 1: Comparison: Atorva 10 mg + EZ vs Atorva 20 mg / Atorva 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, baseline HDL-C, and AVD status; Mean Difference (Final Values) = 3.1, 95% CI [1.5 to 4.8], Standard Error of Mean 0.8 — (Atorva 10 mg + EZ minus Atorva 20 mg / Atorva 40 mg)

9. Other Pre Specified Outcome: Percent Change From Baseline in Non-High Density Lipoprotein Cholesterol (Non-HDL-C) at Week 6
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg
Number analyzed (Participants) | 515 | 515
Percent Change | -23.5 [-25.2 to -21.7] | -11.2 [-13.0 to -9.5]
Statistical Analysis 1: Comparison: Atorva 10 mg + EZ vs Atorva 20 mg / Atorva 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, baseline non-HDL-C, and AVD status; Mean Difference (Final Values) = -12.2, 95% CI [-14.2 to -10.3], Standard Error of Mean 1.0 — (Atorva 10 mg + EZ minus Atorva 20 mg)

10. Other Pre Specified Outcome: Percent Change From Baseline in Non-High Density Lipoprotein Cholesterol (Non-HDL-C) at Week 12
Time Frame: Baseine and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg
Number analyzed (Participants) | 516 | 509
Percent Change | -20.0 [-22.3 to -17.7] | -15.8 [-18.1 to -13.5]
Statistical Analysis 1: Comparison: Atorva 10 mg + EZ vs Atorva 20 mg / Atorva 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, baseline non-HDL-C, and AVD status; Mean Difference (Final Values) = -4.2, 95% CI [-6.8 to -1.7], Standard Error of Mean 1.3 — (Atorva 10 mg + EZ minus Atorva 20 mg)

11. Other Pre Specified Outcome: Percent Change From Baseline in Total Cholesterol (TC) at Week 6
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg
Number analyzed (Participants) | 515 | 516
Percent Change | -15.9 [-17.2 to -14.6] | -8.0 [-9.3 to -6.7]
Statistical Analysis 1: Comparison: Atorva 10 mg + EZ vs Atorva 20 mg / Atorva 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, baseline Total Cholesterol, and AVD status; Mean Difference (Final Values) = -7.9, 95% CI [-9.4 to -6.5], Standard Error of Mean 0.7 — (Atorva 10 mg + EZ minus Atorva 20 mg)

12. Other Pre Specified Outcome: Percent Change From Baseline in Total Cholesterol (TC) at Week 12
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg
Number analyzed (Participants) | 516 | 509
Percent Change | -13.6 [-15.2 to -12.0] | -11.6 [-13.2 to -10.0]
Statistical Analysis 1: Comparison: Atorva 10 mg + EZ vs Atorva 20 mg / Atorva 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, baseline Total Cholesterol, and AVD status; Mean Difference (Final Values) = -2.0, 95% CI [-3.8 to -0.2], Standard Error of Mean 0.9 — (Atorva 10 mg + EZ minus Atorva 20 mg / Atorva 40 mg)

13. Other Pre Specified Outcome: Percent Change From Baseline in Triglycerides (TG) at Week 6
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg
Number analyzed (Participants) | 515 | 516
Percent Change | -12.9 [-14.3 to -9.7] | -5.7 [-8.4 to -3.5]
Statistical Analysis 1: Comparison: Atorva 10 mg + EZ vs Atorva 20 mg / Atorva 40 mg; Test type: Superiority or Other; p < 0.001, Nonparametric ANCOVA; ANCOVA using ranks based on normal scores (Tukey method) with model terms for treatment, baseline TG value (normalized scores), and AVD status; Median Difference (Final Values) = -6.2, 95% CI [-9.0 to -3.4] — (Atorva 10 mg + EZ minus Atorva 20 mg) The median difference is based on the Hodges-Lehmann estimates of shift; The distribution-free 95% CI is based on Wilcoxon's rank sum test statistic

14. Other Pre Specified Outcome: Percent Change From Baseline in Triglycerides (TG) at Week 12
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg
Number analyzed (Participants) | 516 | 509
Percent Change | -11.8 [-13.7 to -9.3] | -8.5 [-11.3 to -7.1]
Statistical Analysis 1: Comparison: Atorva 10 mg + EZ vs Atorva 20 mg / Atorva 40 mg; Test type: Superiority or Other; p < 0.001, Nonparametric ANCOVA; [statistical method as in outcome 13, analysis 1]; Median Difference (Final Values) = -2.1, 95% CI [-5.2 to 1.0] — [estimate comment as in outcome 13, analysis 1]

15. Other Pre Specified Outcome: Percent Change From Baseline in Apo Lipoprotein B (Apo B) at Week 6
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg
Number analyzed (Participants) | 507 | 514
Percent Change | -16.8 [-18.5 to -15.1] | -7.7 [-9.4 to -6.0]
Statistical Analysis 1: Comparison: Atorva 10 mg + EZ vs Atorva 20 mg / Atorva 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, baseline Apo B, and AVD status; Mean Difference (Final Values) = -9.1, 95% CI [-11.0 to -7.3], Standard Error of Mean 0.9 — (Atorva 10 mg + EZ minus Atorva 20 mg)

16. Other Pre Specified Outcome: Percent Change From Baseline in Apo Lipoprotein B (Apo B) at Week 12
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg
Number analyzed (Participants) | 511 | 506
Percent Change | -14.0 [-16.1 to -11.9] | -10.8 [-12.9 to -8.7]
Statistical Analysis 1: Comparison: Atorva 10 mg + EZ vs Atorva 20 mg / Atorva 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, baseline Apo B, and AVD status; Mean Difference (Final Values) = -3.2, 95% CI [-5.5 to -0.9], Standard Error of Mean 1.2 — (Atorva 10 mg + EZ minus Atorva 20 mg / Atorva 40 mg)

17. Other Pre Specified Outcome: Percent Change From Baseline in Apo Lipoprotein A-I (Apo A-I) at Week 6
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg
Number analyzed (Participants) | 507 | 514
Percent Change | -1.1 [-2.4 to 0.3] | -1.7 [-3.0 to -0.3]
Statistical Analysis 1: Comparison: Atorva 10 mg + EZ vs Atorva 20 mg / Atorva 40 mg; Test type: Superiority or Other; p = 0.401, ANCOVA; Model terms: treatment, baseline Apo A-I, and AVD status; Mean Difference (Final Values) = 0.6, 95% CI [-0.9 to 2.1], Standard Error of Mean 0.8 — (Atorva 10 mg + EZ minus Atorva 20 mg)

18. Other Pre Specified Outcome: Percent Change From Baseline in Apo Lipoprotein A-I (Apo A-I) at Week 12
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg
Number analyzed (Participants) | 511 | 506
Percent Change | 0.7 [-0.7 to 2.1] | -2.0 [-3.4 to -0.6]
Statistical Analysis 1: Comparison: Atorva 10 mg + EZ vs Atorva 20 mg / Atorva 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, baseline Apo A-I, and AVD status; Mean Difference (Final Values) = 2.7, 95% CI [1.1 to 4.2], Standard Error of Mean 0.8 — (Atorva 10 mg + EZ minus Atorva 20 mg / Atorva 40 mg)

19. Other Pre Specified Outcome: Percent Change From Baseline in Total Cholesterol (TC): High Density Lipoprotein Cholesterol (HDL-C) Ratio at Week 6
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg
Number analyzed (Participants) | 515 | 515
Percent Change | -16.9 [-18.4 to -15.3] | -7.9 [-9.4 to -6.3]
Statistical Analysis 1: Comparison: Atorva 10 mg + EZ vs Atorva 20 mg / Atorva 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, baseline Total-C:HDL-C, and AVD status; Mean Difference (Final Values) = -9.0, 95% CI [-10.7 to -7.3], Standard Error of Mean 0.9 — (Atorva 10 mg + EZ minus Atorva 20 mg)

20. Other Pre Specified Outcome: Percent Change From Baseline in Total Cholesterol (TC):High Density Lipoprotein Cholesterol (HDL-C) Ratio at Week 12
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg
Number analyzed (Participants) | 516 | 509
Percent Change | -14.4 [-16.4 to -12.5] | -9.8 [-11.8 to -7.9]
Statistical Analysis 1: Comparison: Atorva 10 mg + EZ vs Atorva 20 mg / Atorva 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, baseline Total-C:HDL-C, and AVD status; Mean Difference (Final Values) = -4.6, 95% CI [-6.8 to -2.4], Standard Error of Mean 1.1 — (Atorva 10 mg + EZ minus Atorva 20 mg / Atorva 40 mg)

21. Other Pre Specified Outcome: Percent Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C):High Density Lipoprotein Cholesterol (HDL-C) Ratio at Week 6
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg
Number analyzed (Participants) | 515 | 515
Percent Change | -27.2 [-29.5 to -25.0] | -12.6 [-14.9 to -10.4]
Statistical Analysis 1: Comparison: Atorva 10 mg + EZ vs Atorva 20 mg / Atorva 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, baseline LDL-C:HDL-C, and AVD status; Mean Difference (Final Values) = -14.6, 95% CI [-17.0 to -12.2], Standard Error of Mean 1.2 — (Atorva 10 mg + EZ minus Atorva 20 mg)

22. Other Pre Specified Outcome: Percent Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C):High Density Lipoprotein Cholesterol (HDL-C) Ratio at Week 12
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg
Number analyzed (Participants) | 516 | 509
Percent Change | -22.9 [-25.9 to -20.0] | -16.0 [-18.9 to -13.1]
Statistical Analysis 1: Comparison: Atorva 10 mg + EZ vs Atorva 20 mg / Atorva 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, baseline LDL-C:HDL-C, and AVD status; Mean Difference (Final Values) = -6.9, 95% CI [-10.1 to -3.7], Standard Error of Mean 1.7 — (Atorva 10 mg + EZ minus Atorva 20 mg / Atorva 40 mg)

23. Other Pre Specified Outcome: Percent Change From Baseline in Apo Lipoprotein B (Apo B):Apo Lipoprotein A-I (Apo A-I) Ratio at Week 6
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg
Number analyzed (Participants) | 507 | 514
Percent Change | -14.8 [-16.6 to -12.9] | -5.2 [-7.1 to -3.4]
Statistical Analysis 1: Comparison: Atorva 10 mg + EZ vs Atorva 20 mg / Atorva 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, baseline Apo B:Apo A-I, and AVD status; Mean Difference (Final Values) = -9.5, 95% CI [-11.6 to -7.5], Standard Error of Mean 1.0 — (Atorva 10 mg + EZ minus Atorva 20 mg)

24. Other Pre Specified Outcome: Percent Change From Baseline in Apo Lipoprotein B (Apo B):Apo Lipoprotein A-I (Apo A-I) Ratio at Week 12
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg
Number analyzed (Participants) | 511 | 506
Percent Change | -13.5 [-15.7 to -11.3] | -8.2 [-10.4 to -6.0]
Statistical Analysis 1: Comparison: Atorva 10 mg + EZ vs Atorva 20 mg / Atorva 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, baseline Apo B:Apo A-I, and AVD status; Mean Difference (Final Values) = -5.3, 95% CI [-7.7 to -2.9], Standard Error of Mean 1.2 — (Atorva 10 mg + EZ minus Atorva 20 mg / Atorva 40 mg)

25. Other Pre Specified Outcome: Percent Change From Baseline in Non-High Density Lipoprotein Cholesterol (Non-HDL):High Density Lipoprotein Cholesterol (HDL-C) Ratio at Week 6
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg
Number analyzed (Participants) | 515 | 515
Percent Change | -24.0 [-26.2 to -21.8] | -11.1 [-13.3 to -8.9]
Statistical Analysis 1: Comparison: Atorva 10 mg + EZ vs Atorva 20 mg / Atorva 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, baseline non-HDL-C:HDL-C, and AVD status; Mean Difference (Final Values) = -12.9, 95% CI [-15.3 to -10.5], Standard Error of Mean 1.2 — (Atorva 10 mg + EZ minus Atorva 20 mg)

26. Other Pre Specified Outcome: Percent Change From Baseline in Non-High Density Lipoprotein Cholesterol (Non-HDL):High Density Lipoprotein Cholesterol (HDL-C) Ratio at Week 12
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg
Number analyzed (Participants) | 516 | 509
Percent Change | -20.4 [-23.2 to -17.6] | -13.8 [-16.6 to -10.9]
Statistical Analysis 1: Comparison: Atorva 10 mg + EZ vs Atorva 20 mg / Atorva 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, baseline non-HDL-C:HDL-C, and AVD status; Mean Difference (Final Values) = -6.7, 95% CI [-9.8 to -3.6], Standard Error of Mean 1.6 — (Atorva 10 mg + EZ minus Atorva 20 mg / Atorva 40 mg)

27. Other Pre Specified Outcome: Percent Change From Baseline in Ratio of Highly Selective C-Reactive Protein (Hs-CRP) at Week 6
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg
Number analyzed (Participants) | 497 | 500
Percent Change | -13.5 [-19.6 to -6.8] | -10.7 [-17.0 to -3.9]
Statistical Analysis 1: Comparison: Atorva 10 mg + EZ vs Atorva 20 mg / Atorva 40 mg; Test type: Superiority or Other; p = 0.534, Longitudinal Data Analysis (LDA); LDA method of Liang and Zeger with model terms: treatment, time, AVD status, and the interaction of time by treatment; Mean Difference (Final Values) = -2.8, 95% CI [-11.9 to 6.4] — (Atorva 10 mg + EZ minus Atorva 20 mg) Data for analysis was transformed by the natural log and the difference in geometric mean % change from BL calculated based on the difference in the back-transformed least squares means

28. Other Pre Specified Outcome: Percent Change From Baseline in Ratio of Highly Selective C-Reactive Protein (Hs-CRP) at Week 12
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg
Number analyzed (Participants) | 506 | 500
Percent Change | -21.7 [-27.3 to -15.6] | -14.6 [-20.7 to -8.0]
Statistical Analysis 1: Comparison: Atorva 10 mg + EZ vs Atorva 20 mg / Atorva 40 mg; Test type: Superiority or Other; p = 0.090, Longitudinal Data Analysis (LDA); LDA method of Liang and Zeger with model terms: treatment, time, AVD status, and the interaction of time by treatment; Mean Difference (Final Values) = -7.0, 95% CI [-15.6 to 1.6] — (Atorva 10 mg + EZ minus Atorva 20 mg / Atorva 40 mg) Data for analysis was transformed by the natural log and the difference in geometric mean % change from BL calculated based on the difference in the back-transformed least squares means

ADVERSE EVENTS:
Description: The number of subjects at risk for reported adverse events is based on an All-Patients-as-Treated population, which includes all randomized patients who received at least one dose of double-blind study therapy
Arm/Group | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg
Serious Adverse Events (participants affected / at risk) | 15 | 14
Other Adverse Events (participants affected / at risk) | 46 | 54
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg
Acute myocardial infarction (Cardiac disorders) | 1/526 | 1/525
Angina pectoris (Cardiac disorders) | 1/526 | 2/525
Angina unstable (Cardiac disorders) | 0/526 | 1/525
Coronary artery disease (Cardiac disorders) | 0/526 | 1/525
Coronary artery occlusion (Cardiac disorders) | 1/526 | 0/525
Myocardial infarction (Cardiac disorders) | 1/526 | 1/525
Abdominal discomfort (Gastrointestinal disorders) | 0/526 | 1/525
Appendicitis perforated (Gastrointestinal disorders) | 1/526 | 0/525
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1/526 | 0/525
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1/526 | 0/525
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1/526 | 0/525
Chest pain (General disorders) | 0/526 | 1/525
Death (General disorders) | 1/526 | 0/525
Empyema (Infections and infestations) | 1/526 | 0/525
Gastroenteritis (Infections and infestations) | 0/526 | 1/525
Pneumonia (Infections and infestations) | 1/526 | 0/525
Pneumonia bacterial (Infections and infestations) | 1/526 | 0/525
Pyelonephritis chronic (Infections and infestations) | 1/526 | 0/525
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/526 | 0/525
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/526 | 0/525
Brain stem haemorrhage (Nervous system disorders) | 0/526 | 1/525
Cerebrovascular accident (Nervous system disorders) | 1/526 | 0/525
Dizziness (Nervous system disorders) | 0/526 | 1/525
Dizziness postural (Nervous system disorders) | 0/526 | 1/525
Intracranial aneurysm (Nervous system disorders) | 0/526 | 1/525
Toxic encephalopathy (Nervous system disorders) | 1/526 | 0/525
Transient ischemic attack (Nervous system disorders) | 0/526 | 1/525
Urinary retention (Renal and urinary disorders) | 1/526 | 0/525
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0/526 | 1/525
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0/526 | 1/525
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0/526 | 1/525
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1/526 | 0/525
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1/526 | 0/525
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Atorva 10 mg + EZ | Atorva 20 mg / Atorva 40 mg
Constipation (Gastrointestinal disorders) | 7/526 | 3/525
Bronchitis (Infections and infestations) | 6/526 | 3/525
Nasopharyngitis (Infections and infestations) | 6/526 | 7/525
Upper respiratory tract infection (Infections and infestations) | 7/526 | 8/525
Asparate aminotransferase increased (Investigations) | 2/526 | 5/525
Blood glucose increased (Investigations) | 5/526 | 2/525
Back pain (Musculoskeletal and connective tissue disorders) | 4/526 | 6/525
Muscle spasm (Musculoskeletal and connective tissue disorders) | 0/526 | 5/525
Myalgia (Musculoskeletal and connective tissue disorders) | 5/526 | 4/525
Headache (Nervous system disorders) | 7/526 | 7/525
Hypertension (Vascular disorders) | 0/526 | 9/525

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.